CLINICAL TRIAL: NCT06751329
Title: A Phase I, Multicentre, Open-label, First-in-Human, Dose Escalation and Expansion Study of DM002 in Patients With Advanced Solid Tumors
Brief Title: A Study of DM002 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xadcera Biopharmaceutical (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Doma Biopharmaceutical（Suzhou）Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DM002001
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Neoplasms; Prostatic Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms; Solid Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Prostatic Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Level 1 (Experimental): 1.0 mg/kg
  Interventions: Drug: DM002
- Dose Level 2 (Experimental): ≤2.0 mg/kg
  Interventions: Drug: DM002
- Dose Level 3 (Experimental): ≤3.0 mg/kg,
  Interventions: Drug: DM002
- Dose Level 4 (Experimental): ≤4.5 mg/kg
  Interventions: Drug: DM002
- Dose Level 5 (Experimental): ≤6.0 mg/kg
  Interventions: Drug: DM002
- Dose Level 6 (Experimental): ≤7.5 mg/kg
  Interventions: Drug: DM002

INTERVENTIONS:
Drug: DM002 — An IV infusion of DM002 will be administrated approximately 30-60 min on D1 once Q3W

SUMMARY:
The goal of study：

The study has two parts: Part 1 Dose Escalation and Part 2 Dose Expansion.

In Part 1, a few participants will receive the lowest dose of study drug. The study team will make sure it is safe and tolerated before enrolling new participants at a higher dose of study drug. There will be up to six or more dose levels of study drug tested (called cohorts). Which dose you receive will depend on how many participants have taken part in the study before you.

The purpose of Part 1 of the study is to evaluate the safety of the study drug at different dose levels, to understand what your body does to the study drug, and to find the best dose of study drug in people who have advanced solid tumor cancers.

In Part 2, participants will receive the best dose level that was determined in Part 1 of the study.

The purpose of Part 2 of the study is to evaluate the safety of the study drug at the dose level determined in Part 1, to understand what your body does to the study drug, and to see how your cancer responds to the study drug.

Participants will:

Participants will have 17 or more visits to the study centre. This study has a screening phase of up to 28 days , and a treatment phase with cycles of 21 days each. Participants will also have an End of Treatment (EOT) visit 21 days after the final study drug treatment, and a Follow-up visit 30 days after the EOT visit . Participants will be contacted by telephone every 3 months after the Follow-up visit to check on the wellbeing and record any new anticancer therapy they may have started.

DETAILED DESCRIPTION:
DM002, a bispecific antibody-drug conjugate (ADC) developed using fully human antibodies with a common light chain, which targets MUC1 and HER3.

DM002 is sterile yellowish-green lyophilized powder for intravenous (IV) infusion. Subjects with solid malignant tumors will be treated with DM002 IV on Day 1 once every 3 weeks (Q3W) (dose adjustments may be required depending on the safety profile and PK data of each dose).

ELIGIBILITY:
Inclusion Criteria:

Common Inclusion Criteria (Part 1 and Part 2)

1. Subjects must have the ability to understand and willingness to sign a written informed consent document.
2. Subjects must be ≥18 years of age at the time of signing the informed consent form.
3. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
4. Has a life expectancy of ≥3 months.
5. Participants must meet the following laboratory values within 7 days prior to first dose of study drug:

   Note: Transfusion (red blood cell or platelet) or granulocyte-colony stimulating factor (G-CSF) administration is not allowed within 2 weeks prior to laboratory assessments at Screening.
   * Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L;
   * Platelet count ≥100 × 10⁹/L;
   * Hemoglobin ≥9 g/dL;
   * Calculated creatinine clearance (CrCL) >60 mL/min (Cockroft-Gault Equation);
   * Total bilirubin ≤ 1.5 x ULN;
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 × upper limit of normal (ULN), if liver metastases are present, ≤5 × ULN;
   * International normalized ratio (INR)<2.0, and prothrombin time and either partial thromboplastin time (PTT) or activated PTT (aPTT) ≤1.5 × ULN, except for participants receiving anti-vitamin K derivative anticoagulant therapy who must have prothrombin time/INR within therapeutic range as deemed appropriate by the Investigator.
6. Has measurable disease based on RECIST version 1.1.
7. Participants are required to provide tumor tissue specimens obtained within the previous 3 years for the measurement of MUC1 and/or HER3 and other biomarkers. For those subjects who are unable to provide tissue samples will be encouraged (but not mandatory) to undergo biopsy if the risk is manageable. If the biopsy is not possible, it should inform the sponsor for enrolment.

Exclusion Criteria:

1. Subjects have another active invasive malignancy within 5 years, with the following exceptions and notes:

   1. History of noninvasive malignancy, such as cervical cancer in situ, in situ melanoma, or ductal carcinoma in situ of the breast that is in complete remission 5 years after treatment with curative intent is allowed.
   2. Malignancies with a negligible risk of metastasis or death (such as adequately treated basal or squamous cell skin cancer and localized prostate cancer).
2. Current or history of a hematologic malignancy.
3. Anticancer therapy (chemotherapy, immunotherapy, hormonal therapy, targeted therapy, biologic therapy, or other anti-cancer therapies, except for hormones for hypothyroidism or estrogen replacement therapy, anti-estrogen analogs, agonists required to suppress serum testosterone levels) within 28 days or 5 half-lives, whichever is shorter, prior to the first study dose. Radiotherapy with a wide field of radiation within 28 days, or radiotherapy with a limited field of radiation for palliation within 14 days of the first study dose. Major surgery, other than diagnostic surgery, within 4 weeks of the first study dose.
4. Primary central nervous system (CNS) malignancies or CNS metastases. Individuals with brain metastases can be enrolled only if treated, nonprogressive brain metastases and off high-dose steroids (>20 mg prednisone or equivalent) for at least 4 weeks.
5. History of known allergies to ADC, or prior discontinuation of an ADC due to treatment-related toxicities. Has received prior treatment with ADCs that include topoisomerase I (Topo I) payload, and treatment history with any investigational drug within 4 weeks before enrolment in the study.
6. Has an uncontrolled infection requiring IV injection of antibiotics, antivirals, or antifungals.
7. Has a pre-existing clinically significant lung diseases (e.g., interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis) or pre-existing ocular disorders.
8. Clinically uncontrolled intercurrent illness, including but not limited to an ongoing active infection, active coagulopathy, uncontrolled cardiovascular disease, uncontrolled immune disease, uncontrolled diabetes, uncontrolled pleural and peritoneal effusion, psychiatric illness that would limit compliance with the study requirements and other serious medical illnesses requiring systemic therapies.
9. Mean resting corrected QT interval corrected by Fridericia's formula (QTcF) >470 msec obtained from triplicate 12-lead ECGs at baseline; using concomitant medications that would prolong the QT interval.
10. Left ventricular ejection fraction <50% by either an echocardiogram (ECHO) or a multi-gated acquisition scan within 28 days before first dose of the study drug.
11. Known active hepatitis B (HBV) or hepatitis C (HCV) infection. Chronic carriers of HBV infection (HBsAg-positive, undetectable HBV DNA or HBV DNA ≤2500 copies/ml or 500 IU/ml) receive prophylactic treatment during the study can be enrolled. Participants with a history of HCV infection have completed curative antiviral treatment and HCV viral load below the limit of quantification and HCV antibody positive but HCV ribonucleic acid (RNA) negative due to prior treatment or natural resolution should be eligible.
12. Known human immunodeficiency virus (HIV) infection which is not well controlled. Participants should be tested for HIV prior to enrollment if required by local regulations or institutional review board (IRB)/ethics committee. All the following criteria are required to define an HIV infection (positive HIV1/2 antibodies test) that is well controlled: HIV viral load <400 copies/mL, CD4+ T- cell counts ≥350 cells/μL, no history of acquired immunodeficiency syndrome-defining opportunistic infection within the past 12 months, and stable viral load for at least 4 weeks on same anti-HIV retroviral medications.
13. Subjects who are from endemic areas (refer to WHO high tuberculosis burden country list, China is endemic area) will be specifically screened for tuberculosis with any available test. Subjects with active tuberculosis are excluded. Subjects who have received bacille Calmette-Guerin vaccination may have a false positive result of purified-protein derivative (PPD) test. These subjects are eligible if they have a negative result of interferon gamma release assay (IGRA).
14. Has received a live vaccine within 30 days prior to the first dose of study drug.
15. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia and anemia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, ≤Grade 1 or baseline. Note: Participants may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to enrolment/randomization and managed with the standard treatment) that the Investigator deems related to previous anticancer therapy, following discussion with the Sponsor's medical monitor, such as the following: Grade 2 chemotherapy-induced neuropathy, hypothyroidism, hyperglycemia.
16. Females who are pregnant or lactating or who intend to become pregnant during participation in the study are not eligible to participate.
17. Participants who are of reproductive potential refuse to use effective methods of birth control during participation of the study and within 7 months for female (and 4 months for male) after the last dose administration.
18. Participants who took drugs or food which can strongly inhibit or induce the cytochrome P450 (CYP) isoenzyme, CYP3A4/5 within 2 weeks prior to the first dose of DM002 or within 5 half-lives, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-10-08 (Estimated); Study Completion 2028-04-18 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) of DM002 | 12 months
  Incidence of DLTs of DM002 will be determined. A dose-limiting toxicity (DLT) is defined as grade 3 neurological toxicities (e.g. chemical meningitis) or other grade 4 toxicities.
Maximum tolerated dose (MTD) for DM002 | 12 months
  The MTD of DM002 will be determined. The MTD is defined as the dose where 0/3 or 1/6 patients experienced a DLT with at least two patients encountering DLT at the higher dose.

SECONDARY OUTCOMES:
Area Under the Curve（AUC，ng·h/mL） | 12 months
  Area under the plasma concentration-time curve from time zero extrapolated to infinity, calculated by linear up/log down trapezoidal summation.
Maximum (peak) plasma concentration (Cmax, ng/mL) | 12 months
  Maximum concentration, obtained directly from the observed concentration versus time data.
Time to maximum (peak) concentration (Tmax, h) | 12 months
  Time to Cmax
Trough concentration (Ctrough, ng/mL) | 12 months
  The lowest plasma concentration reached before the next dose.
Objective response rate (ORR) | 12 months
  ORR is defined as the number of patients with at least a confirmed complete response (CR) or partial response (PR), based on the best objective response values while on treatment using RECIST version 1.1

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Scientia Clinical Research, Randwick, New South Wales
  - Cancer Care Wollongong, Wollongong, New South Wales
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia